CLINICAL TRIAL: NCT00379613
Title: A Multi-Center Randomized Safety Assessor-Blinded Placebo-Controlled Parallel and Dose Escalating Dose-Finding Trial in Subjects of ASA 1 - 2 to Assess the Safety, Efficacy and PK of Sugammadex Administered at 5 Min. After Administration of 1.2 mg/kg Esmeron
Brief Title: Use of Sugammadex Administered at 5 Minutes After Administration of 1.2 mg/kg Esmeron® (19.4.205)(P05942)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05942; 19.4.205
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Placebo Comparator): rocuronium + 16.0 mg/kg Org 25969
  Interventions: Drug: Placebo
- 2 (Experimental): rocuronium + 2.0 mg/kg Org 25969
  Interventions: Drug: sugammadex
- 3 (Experimental): rocuronium + 4.0 mg/kg Org 25969
  Interventions: Drug: sugammadex
- 4 (Experimental): rocuronium + 8.0 mg/kg Org 25969
  Interventions: Drug: sugammadex
- 5 (Experimental): rocuronium + 12.0 mg/kg Org 25969
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — After induction of anesthesia an intubation dose of NMBA was administered IV: 1.2 mg/kg rocuronium (arms 2-6)
  At 5 minutes after administration of rocuronium, the randomized single dose of sugammadex 2.0 to 16.0 mg/kg IV was administered
  Other Names: Org 25969
  Arms: 2; 3; 4; 5
Drug: Placebo — After induction of anesthesia an intubation dose of NMBA was administered IV: 1.2 mg/kg rocuronium (arms 2-6)
  At 5 minutes after administration of rocuronium, the randomized single dose of sugammadex 2.0 to 16.0 mg/kg IV was administered
  Arms: 1

SUMMARY:
The purpose of this study is to determine the optimal dose of sugammadex when this compound is administered during deep neuromuscular block. Sugammadex is administered shortly (5 minutes) after administration of a high dose (1.2 mg/kg) of the neuromuscular blocking agent rocuronium . Under these circumstance the neuromuscular block is deep. The safety and pharmacokinetics of sugammadex are also studied.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - 2 between the ages of 18 and 64, inclusive
* Scheduled for surgical procedures with an anticipated duration of anesthesia of at least 90 minutes, without further need for muscle relaxation other than for intubation
* Scheduled for surgery in supine position
* Given written informed consent

Exclusion Criteria:

* Subjects in whom a difficult intubation because of anatomical malformations was expected
* Subjects known or suspected to have neuromuscular disorders impairing neuromuscular block (NMB) and/or significant renal dysfunction
* Subjects known or suspected to have a (family) history of malignant hyperthermia
* Subjects known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia
* Subjects receiving medication known to interfere with neuromuscular blocking agents such as anticonvulsants and Mg2+
* Subjects who had already participated in CT 19.4.205
* Subjects who had participated in another clinical trial, not pre-approved by NV Organon, within 30 days of entering into CT 19.4.205
* Female subjects who are pregnant: in females pregnancy was to be excluded both from medical history and by an hCG test within 24 hours before surgery except in females who were not of childbearing potential i.e. at least 2 years postmenopausal or underwent tubal ligation or an hysterectomy
* Females of childbearing potential not using an acceptable method of birth control: condom or diaphragm with spermicide, vasectomized partner (>6 months), IUD, abstinence
* Subjects giving breast-feeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2003-11-07 (Actual); Primary Completion 2004-07-14 (Actual); Study Completion 2004-07-14 (Actual)

PRIMARY OUTCOMES:
Time from start administration of sugammadex to recovery T4/T1 ratio to 0.9. | After administration of rocuronium

SECONDARY OUTCOMES:
Time from start administration of sugammadex to recovery T4/T1 ratio to 0.7; Time from start administration of sugammadex to recovery T4/T1 ratio to 0.8. | After administration of rocuronium

REFERENCES:
- [Result] de Boer HD, Driessen JJ, Marcus MA, Kerkkamp H, Heeringa M, Klimek M. Reversal of rocuronium-induced (1.2 mg/kg) profound neuromuscular block by sugammadex: a multicenter, dose-finding and safety study. Anesthesiology. 2007 Aug;107(2):239-44. doi: 10.1097/01.anes.0000270722.95764.37. PMID 17667567
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html